CLINICAL TRIAL: NCT07368907
Title: Walk On! National Council on Aging Innovation Lab
Acronym: Walk On! NCOA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Council on Aging (NCOA) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB00138002; 90ACIL0001 (Other Grant/Funding Number: Administration for Community Living/Health and Human Services)
Record Dates: First submitted 2026-01-20; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2025-12

CONDITIONS: Falls Prevention
Keywords: Mobility Limitation; Implementation Science; Community-based
MeSH Terms: conditions — Mobility Limitation

STUDY DESIGN:
Intervention Model Description: This study uses a single-group interventional model in which all participating Community-Based Organizations (CBOs) receive the same implementation support to promote program adoption. All older adult participants enrolled will receive the intervention. All activities will be unblinded. All intervention activities will take place in person within a community setting. Intervention participants will be older adults, including those with mobility limitations, recruited from the local community. The intervention will focus on improving walking endurance, strength, and balance. The intervention will be delivered by trained facilitators based at CBOs. All facilitators will receive comprehensive training and implementation support as part of this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Walk On! Program (Experimental): This study uses a single-group model in which all participating Community-Based Organizations (CBOs) receive the same implementation support for Walk On! intervention adoption and delivery. All older adult participants enrolled will receive the intervention. All activities will be unblinded. Intervention participants will be older adults, including those with mobility limitations, recruited from the local community. All intervention activities will take place in person within a community setting. The intervention will focus on improving walking endurance, strength, and balance. The intervention will be delivered by trained facilitators based at CBOs. All facilitators will receive comprehensive training and implementation support as part of this study.
  Interventions: Behavioral: Walk On! Program

INTERVENTIONS:
Behavioral: Walk On! Program — 24 sessions (twice weekly for 60 minutes over 12 weeks) with a focus on improving walking endurance, strength, and balance in older adults, including those with mobility limitations. All intervention activities will take place in person within a community setting. The intervention will be delivered by trained facilitators based at community-based organizations. All facilitators will receive comprehensive training and implementation support as part of this study.

SUMMARY:
This is a multi-site, one-arm type-2 hybrid-effectiveness implementation trial. The goal of this clinical trial is to learn if the Walk On! program helps prevent falls in older adults who have trouble moving around or feel socially isolated. Researchers want to know:

1. What are the best ways for organizations to offer the Walk On! program and keep it running for older adults in their community?
2. Does Walk On! help prevent falls in older adults?

Older Adult Participants will:

1. Join group walking sessions led by a trained facilitator
2. Meet twice a week for 12 weeks (24 sessions)
3. Take part in simple tests before and after the program to see if there are any changes in older adults' function, confidence in not falling, or loneliness.

DETAILED DESCRIPTION:
Despite the clear benefits of walking for individuals at risk of mobility disability, no National Council on Aging (NCOA)-approved evidence-based health programs emphasize walking in a supervised setting, particularly over longer distances. While some programs offer chair exercise, balance, and yoga/tai chi, these do not focus on structured, progressive walking for older adults with limited mobility. Additionally, many older adults living in rural areas have described living in a "health desert" with limited access to evidence-informed health promotion programs.

Walk On! is designed to provide community-based walking for older adults who are physically, socially and/or geographically isolated. This includes a focus on older adults with existing functional limitations and/or mobility challenges that may otherwise limit one's participation in community-based programs and/or individuals who live in rural areas without easy access to safe walking spaces. An underlying goal of this project is to expand access to Walk On! by starting programs in new spaces and places across diverse service sectors.

In brief, Walk On! is a facilitator-led, group-based program consisting of 24 sessions (twice weekly for 60 minutes over a 12 week period) focused on improving walking endurance, strength, and balance for older adults, including those with mobility limitations. Walk On! program facilitators will receive comprehensive implementation support and training to guide their organization in successfully starting and sustaining a program of their own.

Objectives: The long-term goal is to support unique community-based organizations in adopting and sustaining Walk On!. To support this goal this project will evaluate the following objectives:

Objective 1: Evaluate the effectiveness of comprehensive implementation support on community-based organizations adoption and sustainment of Walk On!.

Objective 2: Evaluate the impact of Walk On! on older adults' physical function, falls efficacy, and self-reported loneliness.

ELIGIBILITY:
Program Older Adult Participants: Inclusion Criteria:

* Age greater than or equal to 60 years
* Able to provide own transportation to the program each week
* No planned extended travel or time away during the 12 week program period
* English speaking with intact verbal and written communication skills
* Free of current fracture
* Able to ambulate independently, with or without an assistive device (i.e., cane or walker)

Program Participants: Exclusion Criteria:

* Serious or unstable medical or psychiatric condition that would prevent participation in research study
* Lack of decision-making capacity
* Participated in an evidence-based falls prevention program within the past 12 months

Community-Based Organizations (CBOs): Inclusion Criteria:

* Age greater than or equal to 18 years
* English speaking

Community-Based Organizations (CBOs): Exclusion Criteria:

* Not interested in offering a Walk On! program
* Unwilling and/or unable to participate in implementation activities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Adoption of Program | Week 12
  Number of community-based organizations that deliver of one full 12-week round of Walk On! to a minimum of 8 participants who have not previously participated in the program. Data Source: community-based organization's site attendance records.
Fall Incidence | baseline
  Number of falls in past 12 weeks (3 months), including number of injurious falls.
  Data Source(s): Self-report, pre- and post-program assessment surveys. Number of Survey Items: 2. Total Score range: open-ended, 0 to no upper limit (higher score indicates more falls).
Fall Incidence | week 12
  Number of falls in past 12 weeks (3 months), including number of injurious falls.
  Data Source(s): Self-report, pre- and post-program assessment surveys. Number of Survey Items: 2. Total Score range: open-ended, 0 to no upper limit (higher score indicates more falls).
Fall self-efficacy | baseline
  Confidence in performing daily activities without falling; fear of falling Data Source(s): Self-report, pre- and post-program assessments (Confidence in performing daily activities without falling; fear of falling) Number of Survey Items: 11 Total Score range: 11 to 44 (higher score indicates more confidence in performing daily activities without falling; less fear of falling)
Fall self-efficacy | week 12
  Confidence in performing daily activities without falling; fear of falling. Data Source(s): Self-report, pre- and post-program assessments (Confidence in performing daily activities without falling; fear of falling).
  Number of Survey Items: 11. Total Score range: 11 to 44 (higher score indicates more confidence in performing daily activities without falling; less fear of falling).

SECONDARY OUTCOMES:
Loneliness | baseline, week 12
  Frequency of feelings of isolation and loneliness (never to always). Data Source(s): Self-report, pre- and post-program assessment surveys. Number of Survey items: 2. Total Score Range: 0 to 8 (higher score indicates higher rating of feelings of loneliness and isolation.
Mobility | baseline, week 12
  Definition: Distance walked. Data Source(s): 6-Minute Walk Test, pre- and post-program assessments. Total score range: 0 to no upper limit (higher score indicates greater distance walked, greater mobility) .

OTHER OUTCOMES:
Sustainment of Program | week 36
  Number of community-based organizations that deliver one or more additional full 12-week round(s) of Walk On! to a minimum of 8 participants. Data source is community-based organization's site attendance records.

CONTACTS AND LOCATIONS:
Overall Officials: Jaime M Hughes, MSW, MPH, PhD, Principal Investigator — Wake Forest University Health Sciences

IPD SHARING:
Plan to Share IPD: No